CLINICAL TRIAL: NCT05986513
Title: Investigating Brain Abnormalities in People With Knee Osteoarthritis Using MRI: a Nociplastic Pain Mechanism Based Assessment
Brief Title: Brain MRI for Knee OA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Dinesh Kumbhare, Scientist, Toronto Rehabilitation Institute
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: OAKneeMRI
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Chronic Pain; Central Sensitisation; Knee Osteoarthritis
Keywords: functional magnetic resonance imaging; diffusion tensor imaging; nociplastic pain
MeSH Terms: conditions — Chronic Pain; Osteoarthritis, Knee; Nociplastic Pain

STUDY DESIGN:
Intervention Model Description: Adults who have been clinically diagnosed with knee osteoarthritis (pain free, localized knee pain, or knee and widespread pain) will all receive the same intervention and study protocol.
Who Masked: Outcomes Assessor
Masking Description: The MRI analysis methods are quantitative and unbiased by convention. Furthermore, they will require the researcher to input the age and sex of the participant and indicate if the participant was a healthy control or experimental to allow for group comparisons, but that will not influence the analyses or outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OA-PF (Active Comparator): Individuals with knee OA without knee or bodily pain. All participants will complete the same study protocol with pre- post-perturbation MRI scans and pain assessment questionnaires, as well as breath samples collected at multiple time points during the study visit.
  Interventions: Behavioral: Cold Pressor Gel Test
- OA-Knee (Experimental): Individuals with knee OA with localized knee pain. All participants will complete the same study protocol with pre- post-perturbation MRI scans and pain assessment questionnaires, as well as breath samples collected at multiple time points during the study visit.
  Interventions: Behavioral: Cold Pressor Gel Test
- OA-Knee+Body (Experimental): Individuals with knee OA with localized knee pain and widespread bodily pain. All participants will complete the same study protocol with pre- post-perturbation MRI scans and pain assessment questionnaires, as well as breath samples collected at multiple time points during the study visit.
  Interventions: Behavioral: Cold Pressor Gel Test

INTERVENTIONS:
Behavioral: Cold Pressor Gel Test — This test will allow the research team to induce a painful sensation in participants in a safe, non-invasive, standardized, and short-lasting manner. The protocol for the cold pressor gel test is simple: participants will place their non-dominant hand in the container of cold water for as long as they can up to a maximum of two minutes. If it becomes too painful or uncomfortable during those two minutes, participants can remove their hand from the container. It should be noted again that this is not a treatment for knee OA or chronic pain and will be used to investigate the effects of acute pain in the brain of individuals with a chronic pain condition.

SUMMARY:
It has been estimated that 300 million people worldwide have osteoarthritis (OA), and this has increased by 97% over the past 25 years. OA is degenerative joint disease that has joint cartilage break down and causes the surrounding bone to change and rub. The pain and loss of mobility experienced by people with knee OA can seriously reduce quality of life, while pain management causes significant healthcare spending. Unfortunately, the pain associated with OA is complex and difficult to treat other than to have a total knee replacement surgery to replace the damaged bone and surrounding tissues with artificial ones. Our research study plans to use advanced magnetic resonance imaging techniques and novel analysis methods to determine if specific parts of the brain are responsible for difficult to describe and diagnose aspects of chronic pain. This study will help us better understand the effects of chronic pain in the brain and the results will help guide future research into new therapeutic options that would focus on relieving the brain dysfunction caused by chronic pain.

DETAILED DESCRIPTION:
Chronic pain and knee osteoarthritis - context and gap

Chronic pain is a debilitating concern that can affect the health, employment, and lifestyle of individuals and puts a tremendous strain on the healthcare system. The prevalence of osteoarthritis (OA) is estimated at over 650 million worldwide, and people with knee OA account for 80% of the total burden (Cui et al. 2020). Globally in 2017, knee OA had a prevalence of 263,086,500 and incidence of 12,888,400 (James et al. 2018). A recent study also found that between 19%-43% of adults 40 years and older had knee OA markers, detected using magnetic resonance imaging (MRI), but were asymptomatic (Culvenor et al. 2019). It is estimated that more than 10 million Canadians will have knee OA by the year 2040 (Bombardier et al. 2011) significantly contributing to OA healthcare costs of 1.45 trillion (Bombardier et al. 2011; Sharif et al. 2017). The severity of pain and its impact on function have been identified by people living with knee OA as two of the most important effects of the disease (Smith et al. 2014), contributing to reduced quality of life (Neogi et al. 2013). Uncontrolled OA joint pain is associated with increased healthcare use, therefore improving pain management for OA in Canada may result in a significant healthcare expenditure savings of up to $488 billion (Bombardier et al. 2011). The pain experience and its associated mechanisms in people with knee OA are known to be complex, with alterations in pain signalling (Fingleton et al. 2015) a major factor in susceptibility to the development of persistent pain (Carlesso et al. 2019). Changes in nervous system sensitization do not necessarily correlate with changes in pain, demonstrating that other factors modulating pain, a top-down process, are at play (Skou et al. 2016; Edwards et la. 2016). Interestingly, between 10-20% of knee OA patients continue to experience intense pain even after a total knee replacement indicating that mechanisms beyond those involving joint structures are likely contributing to a complex pain process (Baker et la. 2007; Lundblad et al. 2008; Rice et al. 2018). In a disease where the joint is viewed as an organ in failure (Loeser et al. 2012), phenotyping is necessary to make sense of the heterogeneity. Specific to knee osteoarthritis (OA), pain is associated with changes in the joint structure due to inflammation (e.g., synovitis)(Dainese et al. 2022) or bone marrow lesions (Aso et al. 2021), but the underlying mechanisms are not fully understood (Gwilym et al. 2008).

Nociceptive, neuropathic, and nociplastic pain

In general, pain of known origin falls under two categories based on the cause: (i) nociceptive: pain caused by damage to a bodily tissue; (ii) neuropathic: pain caused by damage to a nerve or nervous system. However, chronic pain that is present without discernable nociceptive or neuropathic components is classified as nociplastic pain (IASP 2022). A recent study by Kosek et al. (2021) developed a simple scale for nociplastic pain diagnosis for clinical pain assessment based on i) the duration/regionality/type of pain, ii) history of hypersensitivities, iii) comorbidity identification, and iv) evoked pain hypersensitivity (Kosek et al 2021). As a visual representation, the Michigan Body Map (MBM) has been validated as a rapid and reliable tool for patients to identify general bodily regions where they experience chronic pain (Brummett et al. 2016). The MBM is a useful and simple tool to determine if pain is localized (i.e., likely nociceptive or neuropathic pain) or widespread (i.e., likely nociplastic pain)(Brummett et al. 2016). To address the unknown chronic pain mechanisms and pain presenting beyond nociceptive or neuropathic injuries, research has been focused on the theory of central sensitization as a phenomenon of nociplastic pain (Fitzcharles et al. 2021; Walsh 2021). The concept of central sensitization is that dysfunction in the central nervous system results in hypersensitivity to noxious and innocuous stimuli (de Boer et al. 2019; Neblett et al. 2013).

Current methods for nociplastic pain assessment

One method being used to examine nociceptive pain is functional magnetic resonance imaging (fMRI) data to measure the neurologic pain signature (NPS)(Han et al. 2022; Wager et al. 2013). The data collected from fMRIs is the brain's blood-oxygen level dependent (BOLD) signal which is closely connected to neurophysiological activation of the brain, and the signal fluctuates based on diamagnetic properties of deoxygenated blood and changes to blood flow and volume to activated or deactivated parts of the brain (Ogawa et al. 1990). The NPS has been shown to be a robust metric for quantitatively assessing the brain's activation in response to pain (Han et al. 2022; Wager et al. 2013). Based on the NPS, humans have several brain regions with key involvement in nociceptive pain interpretation that have proportionately increased or decreased activity relative to an individual's pain (Wager et al. 2013). The activation pattern of the NPS has been shown to be responsive to different forms of quantitative sensory testing (QST) such as thermal, mechanical (Wager et al. 2013), and electrical perturbations (Choi et al. 2011; Rütgen et al. 2015).

In women with chronic joint pain, there is evidence of cortical thinning related to chronic pain that exceeds that of normal aging, especially in the hippocampus, thalamus, and anterior cingulate cortex (de Kruijf et al. 2016). Within the context of OA, several studies have explored the effects of knee OA on fMRI activation changes (López-Solà et al. 2022; Pujol et al. 2017; Yue et al. 2018; Zunhammer et al. 2018). In summary, the studies indicate the BOLD signal is regionally elevated in patients with knee OA, but can be reduced by non-steroidal anti-inflammatory drugs (López-Solà et al. 2022) and analgesics (Yue et al. 2018). Spreading pain and heightened widespread pain sensitivity with corresponding brain abnormalities are commonly found in patients with knee OA (Pujol et al. 2017), and these pain-related brain abnormalities are distinct from potential psychological biases of placebos (Zunhammer et al. 2018).

To address the challenges of identifying the underlying pain mechanisms and providing patient-focused results, our research group has developed an analysis method for resting state fMRI (rsfMRI) and diffusion tensor imaging (DTI) that applies a personalized analysis. Based on the previous research using the NPS, the investigators expect to find regional brain alterations caused by pain that could improve our understanding of chronic pain that are also unique to each patient with knee OA. With our novel analysis, each patient with knee OA will have their MRI data compared to over 88 age- and sex-matched controls and a Z-scoring methodology can identify and objectively quantify abnormal brain regions. This can be applied as a compliment to clinical pain tests and more standard group-wise MRI analyses such as the NPS and functional networks.

While MRI has been useful in indicating brain regions altered by pain, inflammation and excitotoxicity may be underlying pathophysiologies behind nociplastic pain. A possible mechanistic pathway is that of kynurenine, having been linked to several inflammatory conditions, that can be neuroprotective if metabolized into kynurenic acid but neurotoxic if metabolized into quinolinic acid (Savitz 2020; Schwarcz and Stone 2017). Kynurenine is a metabolite of tryptophan and is detectable peripherally using the 13C-Tryptophan Breath Test (13C-TBT)(Teraishi et al. 2015). Although kynurenine has been researched for depression (Teraishi et al. 2015), there is mechanistic overlap at N-methyl-D-aspartate (NMDA) receptors between chronic pain and depression (Savitz 2020; Teraishi et al. 2015; Brandl et al. 2022). Two metabolomic studies of OA patients found decreased tryptophan concentrations (Abdelrazig et al. 2021; Van Pevenage et al. 2022), thus forming the possibility that the kynurenine pathways may be a useful bioindicator for OA.

Our solution for chronic nociplastic pain assessment

This proposed study will be a quantitative examination of nociplastic pain in patients with knee OA. Therefore, the primary objective for this study is to determine if chronic pain, more specifically chronic nociplastic pain, causes neuroplastic brain alterations. It is hypothesized that people with localized chronic pain (OA-Knee) and widespread chronic pain (OA-Knee+Body) exhibit abnormal brain function (e.g., network connectivity and ROI complexity) and reduced microstructural integrity of brain white matter (e.g., decreased fractional anisotropy), that would also be proportionately associated with pain sensitivity and mental state, in comparison to similarly aged individuals with knee osteoarthritis without chronic pain.

The cohort of participants will be separated into three patient groups: the control group will include participants with knee OA but no pain (Osteoarthritis - pain free (OA-PF)), the first exploratory group would include participants with knee OA with pain at the knee (OA-Knee), and the second exploratory group, indicative of chronic nociplastic pain would include people with knee OA with knee and widespread body pain (OA-Knee+Body). Participants in the OA-Knee+Body group will be representative of chronic pain patients presenting with nociplastic pain based on several clinical pain tests (e.g., Nociplastic pain criteria (Kosek et al. 2021), Michigan Body Map (Brummett et al. 2016), knee and wrist QST). Widespread bodily pain will be determined by identifying pain in >3 body regions on the Michigan Body Map and experiencing pain the knee and wrist pain pressure test. This study is designed to acquire resting state functional MRI (rsfMRI) and diffusion tensor imaging (DTI) MRI data at baseline and after experimentally induced pain (i.e., Cold Pressor Gel Test (Lapotka et al. 2017)), and compare the MRI data to clinical pain test results. The exploratory outcomes are to examine if there neuroinflammatory group differences based on the results of the 13C-TBT data.

Study Design

Study participants will be asked to complete a screening appointment over the phone prior to a data collection visit. Prospective participants will be notified of our study by their rheumatologist (i.e., Dr. Adachi) and will contact Dr. Danielli via email if they are interested in participating. Prospective participants will then contact Dr. Danielli to arrange a phone call to verbally obtain consent and perform the screening questions to determine eligibility. The screening visit will take about 30 minutes with Dr. Danielli. As part of the screening process prospective participants will be asked to complete the Nociplastic Pain Criteria (Kosek et al. 2021), the DSM-V Alcohol Use Disorder questionnaire, provide demographic information (i.e., to have balanced age and sex recruitment), and identify possible MRI contraindications. If someone is eligible to participate, an appointment will be then booked for the data collection study visit. All prospective participants will have been diagnosed with knee OA by their rheumatologist and the screening visit will be done to categorize participants into one of three study groups and efficiently book a data collection visit.

Informed written consent will be obtained in accordance with the World Medical Association Declaration of Helsinki prior to any data collection at the data collection study visit. All participants will receive the same data collection protocols. Depending on the preference of the participants, screening and data will be collected at either the Imaging Research Centre (IRC) at St. Joseph's Healthcare Hamilton or the Joint Department of Medical Imaging (JDMI) at Toronto Western Hospital. The questionnaires (i.e., the Depression Anxiety Stress Scale (DASS42)(Crawford et al. 2003), Intermittent and Constant Osteoarthritis Pain (ICOAP)(Hawker et al. 2008; Hawker et al. 2011), and Brief Pain Inventory (BPI)(Cleeland et al. 1991)), and participants will also have a wrist and knee pressure pain threshold tests; these will take about 15 minutes to complete. The baseline and secondary MRI acquisitions would take about 45 minutes each. Participants will be given 5-10 minutes between MRI scan sessions to take a break and stretch their legs. The data collection study visit will last about 2 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis and radiographic evidence of knee OA (by rheumatologist).
2. For the two experimental groups (Groups OA-Knee and OA-Knee+Body), participants must have experienced chronic pain related to their knee OA (>3 months) on most days of each month.
3. Participants in Group OA-Knee+Body must:

   * Exhibit chronic knee pain and widespread bodily pain at >3 Michigan Body Map regions.
   * Meet the Kosek criteria for nociplastic pain: i) the duration/regionality/type of pain, ii) history of hypersensitivities, iii) comorbidity identification, and iv) evoked pain hypersensitivity [19]
4. Participants must be able to speak and understand English.

Exclusion Criteria:

1. Unable to provide consent (e.g., poor English language skills, etc.)
2. History of liver or kidney disease
3. MRI contraindications:

   * Pacemaker
   * Stent
   * Joint prothesis
   * Implanted devices
   * Claustrophobia
   * Pregnant
   * Permanent piercings
4. Chronic/abusive use of alcohol and/or illicit drugs
5. Previous clinical diagnosis of fibromyalgia, a multisite pain disorder, a systemic inflammatory disorder (e.g., rheumatoid arthritis, myopathy), depression, post-traumatic stress disorder
6. Previous stroke or moderate/severe traumatic brain injury, subarachnoid hemorrhage, or intracranial hemorrhage
7. Use of psychotropic medications
8. Control subjects (Group OA-PF) also cannot have a history of chronic pain or knee pain caused by osteoporosis or osteoarthritis
9. Total knee replacement
10. Pregnant or chance of being pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Group and individual differences at baseline and post-intervention | 2 hours
  The primary objective is to determine if chronic pain, more specifically chronic nociplastic pain, causes neuroplastic brain alterations. It is hypothesized that people with localized chronic pain (OA-Knee) and widespread chronic pain (OA-Knee+Body) would exhibit abnormal brain function (e.g., network connectivity and ROI complexity) and reduced microstructural integrity of brain white matter, that would also be proportionately associated with pain sensitivity and mental state, in comparison to similarly aged individuals with knee osteoarthritis without chronic pain.

SECONDARY OUTCOMES:
Presence of neuroinflammation | 2 hours
  The exploratory objective of this study involves peripherally measuring neuroinflammation using the 13C Tryptophan Breath Test (13C-TBT). This test allows our research team to collect exhaled breath samples at multiple time intervals during the data collection study visit after oral consumption of the L-[1-13C]tryptophan and water solution, which based on the metabolism of the labelled tryptophan is a peripheral bioindicator for the presence of neuroinflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Kumbhare, MD, PhD, Principal Investigator — University Health Network, Toronto; Michael D Noseworthy, PhD, PEng, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - Imaging Research Centre, St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Toronto Rehabilitation Institute, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
The data collected for this study will not be shared with researchers outside of the research team.

REFERENCES:
- [Background] Cui A, Li H, Wang D, Zhong J, Chen Y, Lu H. Global, regional prevalence, incidence and risk factors of knee osteoarthritis in population-based studies. EClinicalMedicine. 2020 Nov 26;29-30:100587. doi: 10.1016/j.eclinm.2020.100587. eCollection 2020 Dec. PMID 34505846
- [Background] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Background] Culvenor AG, Oiestad BE, Hart HF, Stefanik JJ, Guermazi A, Crossley KM. Prevalence of knee osteoarthritis features on magnetic resonance imaging in asymptomatic uninjured adults: a systematic review and meta-analysis. Br J Sports Med. 2019 Oct;53(20):1268-1278. doi: 10.1136/bjsports-2018-099257. Epub 2018 Jun 9. PMID 29886437
- [Background] Sharif B, Kopec JA, Wong H, Anis AH. Distribution and Drivers of Average Direct Cost of Osteoarthritis in Canada From 2003 to 2010. Arthritis Care Res (Hoboken). 2017 Feb;69(2):243-251. doi: 10.1002/acr.22933. PMID 27159532
- [Background] Smith TO, Purdy R, Lister S, Salter C, Fleetcroft R, Conaghan P. Living with osteoarthritis: a systematic review and meta-ethnography. Scand J Rheumatol. 2014;43(6):441-52. doi: 10.3109/03009742.2014.894569. Epub 2014 Jun 2. PMID 24882107
- [Background] Neogi T. The epidemiology and impact of pain in osteoarthritis. Osteoarthritis Cartilage. 2013 Sep;21(9):1145-53. doi: 10.1016/j.joca.2013.03.018. PMID 23973124
- [Background] Fingleton C, Smart K, Moloney N, Fullen BM, Doody C. Pain sensitization in people with knee osteoarthritis: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2015 Jul;23(7):1043-56. doi: 10.1016/j.joca.2015.02.163. Epub 2015 Mar 5. PMID 25749012
- [Background] Carlesso LC, Segal NA, Frey-Law L, Zhang Y, Na L, Nevitt M, Lewis CE, Neogi T. Pain Susceptibility Phenotypes in Those Free of Knee Pain With or at Risk of Knee Osteoarthritis: The Multicenter Osteoarthritis Study. Arthritis Rheumatol. 2019 Apr;71(4):542-549. doi: 10.1002/art.40752. Epub 2019 Feb 7. PMID 30307131
- [Background] Skou ST, Roos EM, Simonsen O, Laursen MB, Rathleff MS, Arendt-Nielsen L, Rasmussen S. The efficacy of non-surgical treatment on pain and sensitization in patients with knee osteoarthritis: a pre-defined ancillary analysis from a randomized controlled trial. Osteoarthritis Cartilage. 2016 Jan;24(1):108-16. doi: 10.1016/j.joca.2015.07.013. Epub 2015 Aug 1. PMID 26241775
- [Background] Edwards RR, Dolman AJ, Martel MO, Finan PH, Lazaridou A, Cornelius M, Wasan AD. Variability in conditioned pain modulation predicts response to NSAID treatment in patients with knee osteoarthritis. BMC Musculoskelet Disord. 2016 Jul 13;17:284. doi: 10.1186/s12891-016-1124-6. PMID 27412526
- [Background] Baker PN, van der Meulen JH, Lewsey J, Gregg PJ; National Joint Registry for England and Wales. The role of pain and function in determining patient satisfaction after total knee replacement. Data from the National Joint Registry for England and Wales. J Bone Joint Surg Br. 2007 Jul;89(7):893-900. doi: 10.1302/0301-620X.89B7.19091. PMID 17673581
- [Background] Lundblad H, Kreicbergs A, Jansson KA. Prediction of persistent pain after total knee replacement for osteoarthritis. J Bone Joint Surg Br. 2008 Feb;90(2):166-71. doi: 10.1302/0301-620X.90B2.19640. PMID 18256082
- [Background] Rice DA, Kluger MT, McNair PJ, Lewis GN, Somogyi AA, Borotkanics R, Barratt DT, Walker M. Persistent postoperative pain after total knee arthroplasty: a prospective cohort study of potential risk factors. Br J Anaesth. 2018 Oct;121(4):804-812. doi: 10.1016/j.bja.2018.05.070. Epub 2018 Jul 18. PMID 30236242
- [Background] Loeser RF, Goldring SR, Scanzello CR, Goldring MB. Osteoarthritis: a disease of the joint as an organ. Arthritis Rheum. 2012 Jun;64(6):1697-707. doi: 10.1002/art.34453. Epub 2012 Mar 5. No abstract available. PMID 22392533
- [Background] Dainese P, Wyngaert KV, De Mits S, Wittoek R, Van Ginckel A, Calders P. Association between knee inflammation and knee pain in patients with knee osteoarthritis: a systematic review. Osteoarthritis Cartilage. 2022 Apr;30(4):516-534. doi: 10.1016/j.joca.2021.12.003. Epub 2021 Dec 27. PMID 34968719
- [Background] Aso K, Shahtaheri SM, McWilliams DF, Walsh DA. Association of subchondral bone marrow lesion localization with weight-bearing pain in people with knee osteoarthritis: data from the Osteoarthritis Initiative. Arthritis Res Ther. 2021 Jan 19;23(1):35. doi: 10.1186/s13075-021-02422-0. PMID 33468243
- [Background] Gwilym SE, Pollard TC, Carr AJ. Understanding pain in osteoarthritis. J Bone Joint Surg Br. 2008 Mar;90(3):280-7. doi: 10.1302/0301-620X.90B3.20167. PMID 18310746
- [Background] Kosek E, Clauw D, Nijs J, Baron R, Gilron I, Harris RE, Mico JA, Rice ASC, Sterling M. Chronic nociplastic pain affecting the musculoskeletal system: clinical criteria and grading system. Pain. 2021 Nov 1;162(11):2629-2634. doi: 10.1097/j.pain.0000000000002324. No abstract available. PMID 33974577
- [Background] Brummett CM, Bakshi RR, Goesling J, Leung D, Moser SE, Zollars JW, Williams DA, Clauw DJ, Hassett AL. Preliminary validation of the Michigan Body Map. Pain. 2016 Jun;157(6):1205-1212. doi: 10.1097/j.pain.0000000000000506. PMID 26835782
- [Background] Fitzcharles MA, Cohen SP, Clauw DJ, Littlejohn G, Usui C, Hauser W. Nociplastic pain: towards an understanding of prevalent pain conditions. Lancet. 2021 May 29;397(10289):2098-2110. doi: 10.1016/S0140-6736(21)00392-5. PMID 34062144
- [Background] Walsh DA. Nociplastic pain: helping to explain disconnect between pain and pathology. Pain. 2021 Nov 1;162(11):2627-2628. doi: 10.1097/j.pain.0000000000002323. No abstract available. PMID 34652319
- [Background] den Boer C, Dries L, Terluin B, van der Wouden JC, Blankenstein AH, van Wilgen CP, Lucassen P, van der Horst HE. Central sensitization in chronic pain and medically unexplained symptom research: A systematic review of definitions, operationalizations and measurement instruments. J Psychosom Res. 2019 Feb;117:32-40. doi: 10.1016/j.jpsychores.2018.12.010. Epub 2018 Dec 25. PMID 30665594
- [Background] Neblett R, Cohen H, Choi Y, Hartzell MM, Williams M, Mayer TG, Gatchel RJ. The Central Sensitization Inventory (CSI): establishing clinically significant values for identifying central sensitivity syndromes in an outpatient chronic pain sample. J Pain. 2013 May;14(5):438-45. doi: 10.1016/j.jpain.2012.11.012. Epub 2013 Mar 13. PMID 23490634
- [Background] Han X, Ashar YK, Kragel P, Petre B, Schelkun V, Atlas LY, Chang LJ, Jepma M, Koban L, Losin EAR, Roy M, Woo CW, Wager TD. Effect sizes and test-retest reliability of the fMRI-based neurologic pain signature. Neuroimage. 2022 Feb 15;247:118844. doi: 10.1016/j.neuroimage.2021.118844. Epub 2021 Dec 20. PMID 34942367
- [Background] Wager TD, Atlas LY, Lindquist MA, Roy M, Woo CW, Kross E. An fMRI-based neurologic signature of physical pain. N Engl J Med. 2013 Apr 11;368(15):1388-97. doi: 10.1056/NEJMoa1204471. PMID 23574118
- [Background] Ogawa S, Lee TM, Nayak AS, Glynn P. Oxygenation-sensitive contrast in magnetic resonance image of rodent brain at high magnetic fields. Magn Reson Med. 1990 Apr;14(1):68-78. doi: 10.1002/mrm.1910140108. PMID 2161986
- [Background] Choi JC, Yi DJ, Han BS, Lee PH, Kim JH, Kim BH. Placebo effects on analgesia related to testosterone and premotor activation. Neuroreport. 2011 Jun 22;22(9):419-23. doi: 10.1097/WNR.0b013e32834601c9. PMID 21546858
- [Background] Rutgen M, Seidel EM, Silani G, Riecansky I, Hummer A, Windischberger C, Petrovic P, Lamm C. Placebo analgesia and its opioidergic regulation suggest that empathy for pain is grounded in self pain. Proc Natl Acad Sci U S A. 2015 Oct 13;112(41):E5638-46. doi: 10.1073/pnas.1511269112. Epub 2015 Sep 28. PMID 26417092
- [Background] de Kruijf M, Bos D, Huygen FJ, Niessen WJ, Tiemeier H, Hofman A, Uitterlinden AG, Vernooij MW, Ikram MA, van Meurs JB. Structural Brain Alterations in Community Dwelling Individuals with Chronic Joint Pain. AJNR Am J Neuroradiol. 2016 Mar;37(3):430-8. doi: 10.3174/ajnr.A4556. Epub 2015 Nov 5. PMID 26542234
- [Background] Lopez-Sola M, Pujol J, Monfort J, Deus J, Blanco-Hinojo L, Harrison BJ, Wager TD. The neurologic pain signature responds to nonsteroidal anti-inflammatory treatment vs placebo in knee osteoarthritis. Pain Rep. 2022 Feb 16;7(2):e986. doi: 10.1097/PR9.0000000000000986. eCollection 2022 Mar-Apr. PMID 35187380
- [Background] Pujol J, Martinez-Vilavella G, Llorente-Onaindia J, Harrison BJ, Lopez-Sola M, Lopez-Ruiz M, Blanco-Hinojo L, Benito P, Deus J, Monfort J. Brain imaging of pain sensitization in patients with knee osteoarthritis. Pain. 2017 Sep;158(9):1831-1838. doi: 10.1097/j.pain.0000000000000985. PMID 28683024
- [Background] Yue Y, Collaku A. Correlation of Pain Reduction with fMRI BOLD Response in Osteoarthritis Patients Treated with Paracetamol: Randomized, Double-Blind, Crossover Clinical Efficacy Study. Pain Med. 2018 Feb 1;19(2):355-367. doi: 10.1093/pm/pnx157. PMID 29025005
- [Background] Zunhammer M, Bingel U, Wager TD; Placebo Imaging Consortium. Placebo Effects on the Neurologic Pain Signature: A Meta-analysis of Individual Participant Functional Magnetic Resonance Imaging Data. JAMA Neurol. 2018 Nov 1;75(11):1321-1330. doi: 10.1001/jamaneurol.2018.2017. PMID 30073258
- [Background] Savitz J. The kynurenine pathway: a finger in every pie. Mol Psychiatry. 2020 Jan;25(1):131-147. doi: 10.1038/s41380-019-0414-4. Epub 2019 Apr 12. PMID 30980044
- [Background] Schwarcz R, Stone TW. The kynurenine pathway and the brain: Challenges, controversies and promises. Neuropharmacology. 2017 Jan;112(Pt B):237-247. doi: 10.1016/j.neuropharm.2016.08.003. Epub 2016 Aug 7. PMID 27511838
- [Background] Teraishi T, Hori H, Sasayama D, Matsuo J, Ogawa S, Ota M, Hattori K, Kajiwara M, Higuchi T, Kunugi H. (13)C-tryptophan breath test detects increased catabolic turnover of tryptophan along the kynurenine pathway in patients with major depressive disorder. Sci Rep. 2015 Nov 3;5:15994. doi: 10.1038/srep15994. PMID 26524975
- [Background] Brandl F, Weise B, Mulej Bratec S, Jassim N, Hoffmann Ayala D, Bertram T, Ploner M, Sorg C. Common and specific large-scale brain changes in major depressive disorder, anxiety disorders, and chronic pain: a transdiagnostic multimodal meta-analysis of structural and functional MRI studies. Neuropsychopharmacology. 2022 Apr;47(5):1071-1080. doi: 10.1038/s41386-022-01271-y. Epub 2022 Jan 20. PMID 35058584
- [Background] Abdelrazig S, Ortori CA, Doherty M, Valdes AM, Chapman V, Barrett DA. Metabolic signatures of osteoarthritis in urine using liquid chromatography-high resolution tandem mass spectrometry. Metabolomics. 2021 Mar 3;17(3):29. doi: 10.1007/s11306-021-01778-3. PMID 33655418
- [Background] Van Pevenage PM, Birchmier JT, June RK. Utilizing metabolomics to identify potential biomarkers and perturbed metabolic pathways in osteoarthritis: A systematic review. Semin Arthritis Rheum. 2023 Apr;59:152163. doi: 10.1016/j.semarthrit.2023.152163. Epub 2023 Jan 13. PMID 36736024
- [Background] Crawford JR, Henry JD. The Depression Anxiety Stress Scales (DASS): normative data and latent structure in a large non-clinical sample. Br J Clin Psychol. 2003 Jun;42(Pt 2):111-31. doi: 10.1348/014466503321903544. PMID 12828802
- [Background] Hawker GA, Davis AM, French MR, Cibere J, Jordan JM, March L, Suarez-Almazor M, Katz JN, Dieppe P. Development and preliminary psychometric testing of a new OA pain measure--an OARSI/OMERACT initiative. Osteoarthritis Cartilage. 2008 Apr;16(4):409-14. doi: 10.1016/j.joca.2007.12.015. PMID 18381179
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Cleeland CS, Ryan K. The Brief Pain Inventory. Pain Res Group. 1991;20:143-147.
- [Background] Lapotka M, Ruz M, Salamanca Ballesteros A, Ocon Hernandez O. Cold pressor gel test: A safe alternative to the cold pressor test in fMRI. Magn Reson Med. 2017 Oct;78(4):1464-1468. doi: 10.1002/mrm.26529. Epub 2016 Oct 25. PMID 27779778
- See also: Bombardier C, Hawker G, Mosher D. (2011) The impact of arthritis in Canada: today and over the next 30 years. The Arthritis Alliance of Canada. — https://www.arthritisalliance.ca/en/initiativesen/impact-of-arthritis
- See also: International Association for the Study of Pain (IASP). IASP Terminology. [Accessed on 30 November 2022]. — http://www.iasp-pain.org/resources/terminology/